CLINICAL TRIAL: NCT00738127
Title: Surgical Techniques for Acute Dorsal Trans-Scaphoid Perilunate Dislocations
Brief Title: Safety Study of Surgical Technique to Treat Acute Dorsal Trans-Scaphoid Perilunate Dislocations
Acronym: ADTPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Xu Zhang / MD, The Second Hospital of Qinhuangdao
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHQ-0808-A
Record Dates: First submitted 2008-08-15; First posted 2008-08-20 (Estimated); Last update posted 2008-08-20 (Estimated); Status verified 2008-08

CONDITIONS: Operative Time; Grip Strength; Pain; Functional Status
Keywords: Acute trans-scaphoid perilunate dislocations; Open reduction and internal fixation; Kirschner-wire; Range of motion
MeSH Terms: conditions — Pain | interventions — Open Fracture Reduction; Fracture Fixation, Internal; Methods

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group I (treatment with our technique) Eighteen patients (18 wrists) were available for long-term follow-up at an average of 47.8 months after surgery. There were 11 men and seven women. Their mean age at the time of surgery was 35.4 years (range, 22 to 56 years). The dominant hand was involved in 12 patients and the nondominant hand, in six.
  Interventions: Procedure: Open reduction and internal fixation
- 2 (Experimental): Group II (treatment with Inoue et al.'s technique) Fifteen patients (15 wrists) were evaluated at an average of 51 months. Nine patients were men and 6 were women. The mean age of the group at the time of surgery was 37.5 years (range, 24 to 58 years). The dominant hand was involved in 10 and nondominant hand, in seven.
  Interventions: Procedure: Open reduction and internal fixation

INTERVENTIONS:
Procedure: Open reduction and internal fixation — Inoue et al.'s technique is most commonly used which required placing three K-wires to immobilize both midcarpal joint and radiocarpal joint. This technique is effective, however, it has some problems. In the study, we improve the surgical technique.
  Other Names: Techniques for Perilunate Dislocations

SUMMARY:
The purpose of this study is to determine a surgical technique is effective in the treatment of acute dorsal trans-scaphoid perilunate dislocations.

DETAILED DESCRIPTION:
Open reduction and internal fixation is an effective method of treating acute trans-scaphoid perilunate dislocations. We study a new surgical technique that allows for early wrist excises postoperatively. We compare this technique to Inoue et al. 's techniques affect the objective and subjective outcomes. We also compared the long-term outcomes of these two procedures performed in similar patient groups.Although both groups had satisfactory results with regard to their pain relief, sufficient grip strength and union of scaphoid fracture, the technique using in group I was more easily and quickly to perform. It allows early postoperative excises and results better functional wrist range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical treatment of acute trans-scaphoid perilunate dislocations
* Must have open reduction and internal fixation

Exclusion Criteria:

* Patients whose age under 18 years
* Associated with severe crush, avulsion, or opened injury

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 801 (Actual)
Dates: Start 1992-10; Primary Completion 2004-06 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
In group I was more easily and quickly to perform. It allows early postoperative excises and results better functional wrist range of motion. | 1992-2004

SECONDARY OUTCOMES:
Both groups had satisfactory results with regard to their pain relief, sufficient grip strength and union of scaphoid fracture. | 1992-2004

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, MD, Study Chair — The Second Hospital of Qinhuangdao
Locations (1):
- The Second Hospital of Qinhuangdao, Qinhuangdao, Hebei, China

REFERENCES:
- [Background] Moneim MS, Hofammann KE 3rd, Omer GE. Transscaphoid perilunate fracture-dislocation. Result of open reduction and pin fixation. Clin Orthop Relat Res. 1984 Nov;(190):227-35. PMID 6386257
- See also: Treatment of trans-scaphoid perilunate dislocations by internal fixation with the Herbert screw — http://www.ncbi.nlm.nih.gov/pubmed/2269835
- See also: Perilunate Dislocations — http://www.wheelessonline.com/ortho/perilunate_dislocations
- See also: Acute Dorsal Trans-scaphoid Perilunate Dislocations: Open Reduction and Internal Fixation — http://www.find-health-articles.com/rec_pub_16609406-acute-dorsal-trans-scaphoid-perilunate-dislocations-open-reduction.htm